CLINICAL TRIAL: NCT01836198
Title: Effects of Potent Inhibition of CYP2C8, CYP2J2, and CYP3A4, Using Gemfibrozil, Ketoconazole, and Clarithromycin as Probes, on the Pharmacokinetics of LY2409021 in Healthy Subjects
Brief Title: The Effect of Gemfibrozil, Ketoconazole and Clarithromycin on the Amount of LY2409021 in the Bloodstream
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 14586; I1R-MC-GLBZ (Other: Eli Lilly and Company)
Record Dates: First submitted 2013-04-16; First posted 2013-04-19 (Estimated); Results first posted 2019-03-08 (Actual); Last update posted 2019-03-08 (Actual); Status verified 2018-11

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — adomeglivant; Gemfibrozil; Ketoconazole; Clarithromycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- LY2409021 Only (Part A, Cohort 1) (Experimental): Part A, Period 1. Participants will receive a single 20-milligram (mg) oral dose of LY2409021 on Day 1.
  Interventions: Drug: LY2409021
- LY2409021+Gemfibrozil (Part A, Cohort 1) (Experimental): Part A, Period 2. Participants will receive a morning (AM) and evening (PM) oral dose of 600 mg gemfibrozil on Days 1-20 and an AM oral dose only of 600 mg gemfibrozil on Day 21. Participants will also receive a single 20-mg oral dose of LY2409021 on Day 4.
  Interventions: Drug: LY2409021; Drug: Gemfibrozil
- LY2409021 Only (Part A, Cohort 2) (Experimental): Part A, Period 1. Participants will receive a single 20-mg oral dose of LY2409021 on Day 1.
  Interventions: Drug: LY2409021
- LY2409021+Ketoconazole (Part A, Cohort 2) (Experimental): Part A, Period 2. Participants will receive a once-daily 400-mg oral dose of ketoconazole on Days 1-21 and a single 20-mg oral dose of LY2409021 on Day 4.
  Interventions: Drug: LY2409021; Drug: Ketoconazole
- LY2409021+Clarithromycin (Part B) (Experimental): Part B. Participants will receive a twice-daily 500-mg oral dose of clarithromycin on Days 1-21 and a single 20-mg oral dose of LY2409021 on Day 4.
  Interventions: Drug: LY2409021; Drug: Clarithromycin

INTERVENTIONS:
Drug: LY2409021
Drug: Gemfibrozil
  Arms: LY2409021+Gemfibrozil (Part A, Cohort 1)
Drug: Ketoconazole
  Arms: LY2409021+Ketoconazole (Part A, Cohort 2)
Drug: Clarithromycin
  Arms: LY2409021+Clarithromycin (Part B)

SUMMARY:
The purpose of this study is to examine the effect of gemfibrozil, ketoconazole, and clarithromycin on how much LY2409021 is found in the bloodstream and how long the body takes to get rid of it. The study is split into two parts, Part A and Part B. Participants in Part A are divided into two cohorts (groups). Each cohort will participate in two study periods. Period 1 involves a single dose of LY2409021. Period 2 involves either gemfibrozil or ketoconazole given daily for 21 days with LY2409021 given once on Day 4. Part A will last for 51 days and will also involve screening within 27 days of the start of the study. Part B is only open to participants who successfully completed Part A of the study. Participants in Part B will receive clarithromycin given daily for 21 days with LY2409021 given once on Day 4. Part B will last for 29 days and will also involve screening within 27 days of the start of the study.

DETAILED DESCRIPTION:
Part B was added to the trial in August 2013, per protocol amendment.

ELIGIBILITY:
Inclusion Criteria:

* Participants are overtly healthy males or females, as determined by medical history and physical examination
* Participants have a body mass index (BMI) of 18.0 to 32.0 kilograms per meter squared (kg/m^2), inclusive, at screening
* Participants have a fasting blood glucose of 54 to 110 milligrams per deciliter (mg/dL) (3.0 to 6.1 micromoles per liter [mmol/L])

Exclusion Criteria:

* Participants that have a contraindication to use of clarithromycin
* Participants that have a personal or family history of long QT syndrome
* Participants with a family history of sudden unexplained death or cardiac death in an immediate family member under 60 years of age
* Participants with a personal history of unexplained syncope within the last year
* Participants who have taken drugs or substances known to be an inducer or inhibitor of cytochrome P450 (CYP)3A4 or CYP2C8 or CYP2J2 (for example, St. John's wort, rifampin, ketoconazole, trimethoprim) within 30 days prior to the first dose

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-05; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Evansville, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study was conducted in 2 parts at a single center as an inpatient and outpatient study. Part A was an open-label, fixed sequence, 2-period, 2-cohort study. Part B was an open-label, 1-period study. Participants who completed Part A were eligible to participate in Part B.
Groups:
- Part A: LY2409021+Gemfibrozil (Cohort 1): Part A, Period 1. Participants received a single 20-milligram (mg) oral dose of LY2409021 on Day 1.
  Part A, Period 2. Participants received a morning (AM) and evening (PM) oral dose of 600 mg gemfibrozil on Days 1-20 and an AM oral dose only of 600 mg gemfibrozil on Day 21. Participants also received a single 20-mg oral dose of LY2409021 on Day 4. There was a washout period from Day 22 through Day 28.
- Part A: LY2409021+Ketoconazole (Cohort 2): Part A, Period 1. Participants received a single 20-mg oral dose of LY2409021 on Day 1.
  Part A, Period 2. Participants received a once-daily 400-mg oral dose of ketoconazole on Days 1-21 and a single 20-mg oral dose of LY2409021 on Day 4. There was a washout period from Day 22 through Day 28.
- Part B: LY2409021+Clarithromycin: Part B. Participants received a twice-daily 500-mg oral dose of clarithromycin on Days 1-21 and a single 20-mg oral dose of LY2409021 on Day 4.
Period: Part A, Period 1
Arm/Group | Part A: LY2409021+Gemfibrozil (Cohort 1) | Part A: LY2409021+Ketoconazole (Cohort 2) | Part B: LY2409021+Clarithromycin
Started | 15 | 15 | 0
Received at Least 1 Dose of Study Drug | 15 | 15 | 0
Completed | 15 | 15 | 0
Not Completed | 0 | 0 | 0
Period: Part A, Period 2
Arm/Group | Part A: LY2409021+Gemfibrozil (Cohort 1) | Part A: LY2409021+Ketoconazole (Cohort 2) | Part B: LY2409021+Clarithromycin
Started | 15 | 15 | 0
Completed Part A, Entered Part B | 6 | 6 | 0
Completed | 15 | 14 | 0
Not Completed | 0 | 1 | 0
Not completed — Protocol Violation | 0 | 1 | 0
Period: Part B
Arm/Group | Part A: LY2409021+Gemfibrozil (Cohort 1) | Part A: LY2409021+Ketoconazole (Cohort 2) | Part B: LY2409021+Clarithromycin
Started | 0 | 0 | 12
Received at Least 1 Dose of Study Drug | 0 | 0 | 12
Completed | 0 | 0 | 12
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants enrolled in the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part A: LY2409021+Gemfibrozil (Cohort 1) | Part A: LY2409021+Ketoconazole (Cohort 2) | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.7 (10.8) | 39.5 (11.6) | 39.1 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 15 | 15 | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 15 | 15 | 30
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 6 | 13
  White | 8 | 9 | 17
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics: Area Under the Concentration Curve From Zero to Infinity (AUC[0-∞]) of LY2409021
Time Frame: Predose and 0.5, 1, 2, 4, 8, 12, 24, 48, 72, 96, 144, 216, and 336 hours postdose (and 408, 504, and 576 hours postdose in Part A, Period 2 and Part B only)
Population: All participants who received at least 1 dose of study drug and had evaluable AUC(0-∞) data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hours per milliliter (ng*h/mL)
Groups:
- LY2409021 Only (Part A, Cohort 1); LY2409021 Only (Part A, Cohort 2): Part A, Period 1. Participants received a single 20-mg oral dose of LY2409021 on Day 1.
- LY2409021+Gemfibrozil (Part A, Cohort 1): Part A, Period 2. Participants received a morning (AM) and evening (PM) oral dose of 600 mg gemfibrozil on Days 1-20 and an AM oral dose only of 600 mg gemfibrozil on Day 21. Participants also received a single 20-mg oral dose of LY2409021 on Day 4.
- LY2409021+Ketoconazole (Part A, Cohort 2): Part A, Period 2. Participants received a once-daily 400-mg oral dose of ketoconazole on Days 1-21 and a single 20-mg oral dose of LY2409021 on Day 4.
- LY2409021 Only (Part B Participants, Data From Part A): LY2409021 alone data are from Part A for the participants who participated in Part B.
  Part A, Period 1. Participants received a single 20-mg oral dose of LY2409021 on Day 1.
- LY2409021+Clarithromycin (Part B): Part B. Participants received a twice-daily 500-mg oral dose of clarithromycin on Days 1-21 and a single 20-mg oral dose of LY2409021 on Day 4.
Arm/Group | LY2409021 Only (Part A, Cohort 1) | LY2409021+Gemfibrozil (Part A, Cohort 1) | LY2409021 Only (Part A, Cohort 2) | LY2409021+Ketoconazole (Part A, Cohort 2) | LY2409021 Only (Part B Participants, Data From Part A) | LY2409021+Clarithromycin (Part B)
Number analyzed (Participants) | 15 | 15 | 15 | 14 | 12 | 12
nanogram*hours per milliliter (ng*h/mL) | 34700 (31) | 35300 (35) | 38000 (21) | 145000 (23) | 37400 (25) | 43900 (28)

2. Primary Outcome: Pharmacokinetics: Maximum Concentration (Cmax) of LY2409021
Time Frame: as for outcome 1
Population: All participants who received at least 1 dose of study drug and had evaluable Cmax data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Arm/Group | LY2409021 Only (Part A, Cohort 1) | LY2409021+Gemfibrozil (Part A, Cohort 1) | LY2409021 Only (Part A, Cohort 2) | LY2409021+Ketoconazole (Part A, Cohort 2) | LY2409021 Only (Part B Participants, Data From Part A) | LY2409021+Clarithromycin (Part B)
Number analyzed (Participants) | 15 | 15 | 15 | 15 | 12 | 12
nanograms per milliliter (ng/mL) | 431 (23) | 410 (18) | 445 (19) | 471 (19) | 419 (24) | 467 (23)

ADVERSE EVENTS:
Groups:
- Gemfibrozil Only (Part A, Cohort 1): Part A, Period 2, Days -1 to 3. Participants received a morning (AM) and evening (PM) oral dose of 600 mg gemfibrozil on Days 1-3.
- LY2409021+Gemfibrozil (Part A, Cohort 1): Part A, Period 2, Day 4 to end of Period 2. Participants received a morning (AM) and evening (PM) oral dose of 600 mg gemfibrozil on Days 4-20 and an AM oral dose only of 600 mg gemfibrozil on Day 21. Participants also received a single 20-mg oral dose of LY2409021 on Day 4.
- Ketoconazole Only (Part A, Cohort 2): Part A, Period 2, Days -1 to 3. Participants received a once-daily 400-mg oral dose of ketoconazole on Days 1-3.
- LY2409021+Ketoconazole (Part A, Cohort 2): Part A, Period 2, Day 4 to end of Period 2. Participants received a once-daily 400-mg oral dose of ketoconazole on Days 4-21 and a single 20-mg oral dose of LY2409021 on Day 4.
- Clarithromycin Only (Part B): Part B, Days -1 to 3. Participants received a twice-daily 500-mg oral dose of clarithromycin on Days 1-3.
- LY2409021+Clarithromycin (Part B): Part B, Day 4 to end of Part B. Participants received a twice-daily 500-mg oral dose of clarithromycin on Days 4-21 and a single 20-mg oral dose of LY2409021 on Day 4.
Arm/Group | LY2409021 Only (Part A, Cohort 1) | Gemfibrozil Only (Part A, Cohort 1) | LY2409021+Gemfibrozil (Part A, Cohort 1) | LY2409021 Only (Part A, Cohort 2) | Ketoconazole Only (Part A, Cohort 2) | LY2409021+Ketoconazole (Part A, Cohort 2) | Clarithromycin Only (Part B) | LY2409021+Clarithromycin (Part B)
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/15 | 0/15 | 0/15 | 0/15 | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 6/15 | 1/15 | 5/15 | 5/15 | 2/15 | 9/15 | 1/12 | 8/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LY2409021 Only (Part A, Cohort 1) (N=15) | Gemfibrozil Only (Part A, Cohort 1) (N=15) | LY2409021+Gemfibrozil (Part A, Cohort 1) (N=15) | LY2409021 Only (Part A, Cohort 2) (N=15) | Ketoconazole Only (Part A, Cohort 2) (N=15) | LY2409021+Ketoconazole (Part A, Cohort 2) (N=15) | Clarithromycin Only (Part B) (N=12) | LY2409021+Clarithromycin (Part B) (N=12)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eye irritation (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chapped lips (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Burns second degree (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Excoriation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Foreign body (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Increased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Piloerection (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days